CLINICAL TRIAL: NCT06142305
Title: Ipsilateral Supracondylar Femoral Insufficiency Fractures After Cast Removal of Developmental Dysplasia of the Hip Surgery
Brief Title: Supracondylar Femur Fracture After DDH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hesham Mohamed Elbaseet, Dr., Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCFDDH
Record Dates: First submitted 2023-11-16; First posted 2023-11-21 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: DDH
Keywords: DDH; insufficiency fractures
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Intervention Model Description: incidence of ipsilateral Supracondylar femoral fractures after cast removal for Developmental dysplasia of the hip (DDH) surgery
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DDH surgery (Experimental): DDH surgery open reduction and casting
  Interventions: Procedure: DDH surgery and casting

INTERVENTIONS:
Procedure: DDH surgery and casting — DDH surgery and casting

SUMMARY:
incidence of ipsilateral Supracondylar femoral fractures after cast removal for Developmental dysplasia of the hip (DDH) surgery

ELIGIBILITY:
Inclusion Criteria:

* Age 1-7 years old
* Primary DDH

Exclusion Criteria:

* • Paralytic hip DX in cases of (Cerebral palsy,Meningomyelocele,Neuropathy or Myopathy)

  * Recurrent cases of DDH
  * Past history of ipsilateral distal femoral fractures

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with supracondylar femoral fracture | 6 months
  Number of patients with supracondylar femoral fracture

IPD SHARING:
Plan to Share IPD: No
not planning to share individual participant data (IPD)

REFERENCES:
- [Background] Clinical practice guideline: early detection of developmental dysplasia of the hip. Committee on Quality Improvement, Subcommittee on Developmental Dysplasia of the Hip. American Academy of Pediatrics. Pediatrics. 2000 Apr;105(4 Pt 1):896-905. doi: 10.1542/peds.105.4.896. PMID 10742345